CLINICAL TRIAL: NCT02139813
Title: Prospective Multicentric Randomized Trial of Efficiency and Safety of Laparoscopic Omega Loop Bypass Versus Roux-en-Y Gastric Bypass
Brief Title: Omega Loop Versus Roux-en-Y Gastric Bypass
Acronym: YOMEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014.851
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: Obesity -; Bariatric surgery; Gastric bypass
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Omega Loop Bypass (Experimental): Laparoscopic Mini-gastric bypass
  Interventions: Procedure: Laparoscopic Mini-gastric bypass
- Laparoscopic Roux-en-Y Gastric ByPass (Active Comparator): Procedure of reference in bariatric surgery
  Interventions: Procedure: Procedure of reference in bariatric surgery

INTERVENTIONS:
Procedure: Laparoscopic Mini-gastric bypass — The laparoscopic Omega Loop Bypass will consist of:
  * a long gastric tube, stapled approximately 1.5 cm from the left of the lesser curvature of the antrum to the angle of His
  * a narrow gastric tube will be calibrated to be approximately 1.5 cm wide
  * an Omega loop of 200 cm
  * a unique gastro-jejunal anatomosis of 200cm from the ligament of Treitz, using a linear stapler
  Arms: Laparoscopic Omega Loop Bypass
Procedure: Procedure of reference in bariatric surgery — The laparoscopic Roux-en-Y Gastric Bypass will consist of:
  * a small gastric pouch (about 30cc)
  * an antecolic alimentary limb
  * a gastro-jejunal anastomosis using a linear stapler
  * a 150cm long alimentary limb
  * a 50cm biliary limb
  * a latero-lateral jejuno-jejunal anastomosis
  * closure of the mesenteric defects
  Arms: Laparoscopic Roux-en-Y Gastric ByPass

SUMMARY:
Several prospective trials and metaanalysis have demonstrated the superiority of bariatric surgery on the medical treatment of obesity. The Roux-en-Y Gastric ByPass (RYGBP) procedure has been practiced for more than 30 years, and is the procedure of choice for morbidly obese with metabolic disorders in most of the reference centers. Nevertheless, the RYGBP is a technically demanding procedure with a learning curve of more than 75 cases. The complication rate is around 10% in expert centers.

More recently another procedure has been described which seems as efficient on weight loss and co-morbidities as the RYGBP, with the advantage of being less technically difficult and less morbid, especially for multi-complicated obese and/or the super obese. It consists of a unique gastro-jejunal anastomosis between a long gastric pouch and a jejunal Omega loop. However, this procedure could be at risk of biliary reflux and anastomotic ulcers with dysplastic changes of the gastric and esophageal mucosa. As a result, the Omega loop bypass (OLB) has only been developed by a few teams and remains a controversial subject, particularly as only one monocentric randomized trial has compared it to the RYGBP, which is remains the gold standard. The first litterature results show similar or even better weight loss efficiency than RYGBP with a better feasibility. The early complication rate seems lower, but there are still insufficient data on long term morbidity and biliary reflux consequences.

By performing a randomized and prospective comparison of OLB to RYGBP, the aim of the investigators study is to analyze the weight loss efficiency, the morbidity and mortality, the feasibility, and the quality of life of both techniques, in order to validate the Omega loop bypass as a procedure of choice in bariatric surgery

Hypothesis :

The OLB, while being as efficient as RYGBP on weight loss and metabolic complications, could be less morbid.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old
* Morbid obesity with BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 associated with one or more co-morbidities (type 2 diabetes, arterial hypertension, sleep apnea, dyslipidemia, arthritis)
* Patient who has benefited from an upper GI endoscopy with biopsies
* Patient who has benefited from a pluridisciplinary evaluation, with a favorable opinion for a gastric bypass
* Patient who understands and accepts the need for a long term follow-up
* Patient who agrees to be included in the study and who signs the informed consent form
* Patient affiliated to a healthcare insurance plan

Exclusion Criteria:

* History of esophagitis on upper GI endoscopy (Los Angeles classification)
* Severe gastroesophageal reflux disease (GERD), resistant to medical treatment
* Presence of dysplastic modifications of the gastric mucosa or a history of gastric cancer, on upper gastrointestinal endoscopy.
* Presence of Helicobacter Pylori resistant to medical treatment
* Presence of an unhealed gastro-duodenal ulcer or an ulcer diagnosed less than 2 months previously
* History of previous bariatric surgery (gastric band, sleeve gastrectomy, vertical banded gastroplasty)
* Presence of a severe and evolutive life threatening pathology, unrelated to obesity
* Presence of chronic diarrhea (≥ 3 loose or liquid stools per day, over a period of more than 4 weeks)
* Pregnancy or desire to be pregnant during the study
* Binge eating disorders or other eating disorders according to DSM V criteria
* Mentally unbalanced patients, under supervision or guardianship
* Patient who does not understand French/is unable to give consent
* Patient not affiliated to a French or European healthcare insurance
* Patient who has already been included in a trial which has a conflict of interests with the present study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Weight loss assessment according to Excess BMI Loss percentage (EBL%) | 2 years after surgery
  Weight loss assessment according to Excess BMI Loss percentage (EBL%), calculated using the following formula:
  ((BMI 2 years after surgery - initial BMI) / (initial BMI - 22.5)) X 100

SECONDARY OUTCOMES:
Weight loss according to absolute weight loss (aWL in kg), Excess Weight Loss percentage (EWL%), EBL% | 1, 3, 6, 12, 18 and 24 months after surgery
Waist size reduction according to absolute waist size (in cm) | 1, 3, 6, 12, 18 and 24 months after surgery
Medical and surgical complication rates | 1, 12 and 24 months after surgery
  Medical and surgical complication rates (anastomotic leaks, biliary reflux, bowel obstruction, anastomotic ulcers, anastomotic stenosis, internal hernia, chronic gastritis, esophagitis, iron deficiency anemia …)
Type and severity of complications | During the month following surgery (for early complications) and from one month to 24 months postoperatively (for late complications)
  Type and severity of early and late complications for each procedure, according to the Dindo-Clavien classification
Operative time | Recorded on the day of surgery (Day 0)
  Operative time (expressed in minutes)
Mean length of stay | Average period of 5 days from surgery (Day of surgery = D0) until the end of hospitalization, recorded on Visit 4 (Month1 +/- 10 days)
  Mean length of stay based on the number of days of hospitalization from surgery (Day of surgery = D0) until the end of hospitalization
Patient's quality of life | The day before surgery (D-1) and 6, 12 and 24 months after surgery
  Patient's quality of life score according to the IWQOL questionnaire and the BAROS questionnaire adapted to bariatric surgery
Metabolic and lipid profile | During the period of inclusion (D-60 to D-2) and at 6, 12 and 24 months after surgery
  Metabolic profile of glucose homeostasis and the lipid profile according to antidiabetic and anitilipidemic treatments, HbA1c level, fasting glycemia, HDL, LDL and TG.
Dumping syndrome and hypoglycemia symptoms | At 1, 3,6,12,18 and 24 months after surgery
  Dumping syndrome and hypoglycemia symptoms will be assessed using the Sigstad questionnaire
Gastroesophageal reflux | The day before surgery (Day-1) and 6, 12, and 24 months after surgery
  Gastroesophageal reflux assessed by items 5 and 27 of the GIQLI questionnaire
Modifications of the gastric and esophageal mucosa | 2 years after surgery
  Histological modifications of the gastric and esophageal mucosa, based on upper GI endoscopy with biopsies
Frequency of diarrhea | The day before surgery (day-1) and 6, 12, and 24 months after surgery
  Frequency of diarrhea based on items 7, 30, 31 and 36 of the GIQLI questionnaire
Nutritional status | During the period of inclusion (D-60 to D-2) and 6, 12, and 24 months after surgery (The 24-hour steatorrhea will be quantified at 6 months).
  Nutritional status, assessed by PTH, vitamin B1, B9, B12, and D levels before and 12 and 24 months after surgery and assessed by hemoglobin, albumin, prealbumin, ferritin, saturation coefficient, before and 6, 12 and 24 months after surgery .

CONTACTS AND LOCATIONS:
Overall Officials: Maud ROBERT, MD, Principal Investigator — Service de Chirurgie Digestive - Hôpital Edouard Herriot - Hospices Civils de Lyon - France
Locations (9):
- France (9):
  - Clinique Universitaire de Chirurgie Digestive et de l'Urgence - CHU de Grenoble, Grenoble
  - Cabinet de chirurgie générale, digestive et de l'obésité - Hôpital Privé Drôme et Ardèche, Guilherand-Granges
  - Service de Chirurgie Générale et Endocrinienne - Hôpital Claude Huriez - CHU de Lille, Lille
  - Service de Chirurgie Digestive - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Service de Chirurgie Digestive et Hépato-Bilio-Pancréatique et Transplantation Hépatique - Hôpital de la Pitié Salpêtrière, Paris
  - Service de Chirurgie Digestive, Générale et Cancérologique - Hôpital Européen Georges Pompidou - APHP, Paris
  - Service de Chirurgie Générale - Hôpital Privé de la Loire, Saint-Etienne
  - Service de Chirurgie Générale, Digestive et Viscérale - Centre Hospitalier Intercommunal de Poissy / Saint Gerrmain en Laye, Saint-Germain-en-Laye
  - Service de Chirurgie Digestive et Hépato-Biliaire-Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire

REFERENCES:
- [Result] Robert M, Espalieu P, Pelascini E, Caiazzo R, Sterkers A, Khamphommala L, Poghosyan T, Chevallier JM, Malherbe V, Chouillard E, Reche F, Torcivia A, Maucort-Boulch D, Bin-Dorel S, Langlois-Jacques C, Delaunay D, Pattou F, Disse E. Efficacy and safety of one anastomosis gastric bypass versus Roux-en-Y gastric bypass for obesity (YOMEGA): a multicentre, randomised, open-label, non-inferiority trial. Lancet. 2019 Mar 30;393(10178):1299-1309. doi: 10.1016/S0140-6736(19)30475-1. Epub 2019 Mar 6. PMID 30851879
- [Derived] Robert M, Poghosyan T, Maucort-Boulch D, Filippello A, Caiazzo R, Sterkers A, Khamphommala L, Reche F, Malherbe V, Torcivia A, Saber T, Delaunay D, Langlois-Jacques C, Suffisseau A, Bin S, Disse E, Pattou F. Efficacy and safety of one anastomosis gastric bypass versus Roux-en-Y gastric bypass at 5 years (YOMEGA): a prospective, open-label, non-inferiority, randomised extension study. Lancet Diabetes Endocrinol. 2024 Apr;12(4):267-276. doi: 10.1016/S2213-8587(24)00035-4. Epub 2024 Mar 4. PMID 38452784